CLINICAL TRIAL: NCT05023824
Title: A Prospective, Randomized, Open Label, Parallel Trial Comparing the Efficacy of α-blocker or 5-ARI Withdrawal to Continued Combination Therapy on the Maintenance of LUTS in Men With Benign Prostatic Hyperplasia
Brief Title: Efficacy of α-blocker or 5-ARI Withdrawal to Continued Combination Therapy on the Maintenance of LUTS in Men With BPH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Kyo Chul Koo, Associate Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3-2020-0451; 3-2020-0451 (Other Grant/Funding Number: Handok Pharmaceutical)
Record Dates: First submitted 2021-08-15; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Prostatic Hyperplasia; Prostate Hyperplasia; Prostatic Hypertrophy
Keywords: alpha-blocker; 5α reductase inhibitor; withdrawal; benign prostatic hyperplasia; combination therapy
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Adrenergic alpha-Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- alpha-blocker withdrawal (Experimental): receives 5-ARI monotherapy
  Interventions: Drug: alpha-blocker or 5-ARI withdrawal
- 5-ARI withdrawal (Experimental): receives alpha-blocker monotherapy
  Interventions: Drug: alpha-blocker or 5-ARI withdrawal
- combination therapy (Active Comparator): receives alpha-blocker and 5-ARI
  Interventions: Drug: Maintenance of alpha-blocker and 5-ARI

INTERVENTIONS:
Drug: alpha-blocker or 5-ARI withdrawal — Withdrawal of either alpha-blocker or 5-ARI
  Other Names: alpha-blocker withdrawal; 5-ARI withdrawal
  Arms: 5-ARI withdrawal; alpha-blocker withdrawal
Drug: Maintenance of alpha-blocker and 5-ARI — Maintenance of alpha-blocker and 5-ARI
  Arms: combination therapy

SUMMARY:
The investigators compare the efficacy of alpha-blocker and 5-ARI withdrawal to continued combination therapy on the maintenance of LUTS and improvement of quality of life outcomes in men with benign prostatic hyperplasia.

DETAILED DESCRIPTION:
Benign Prostatic Hyperplasia (BPH) is the primary cause of lower urinary tract symptoms (LUTS). Combination therapy with an alpha-blocker and 5α reductase inhibitors (5-ARI) is the first-line treatment of BPH-related LUTS for the reduction of the size of the prostate and LUTS improvement. Combination therapy is tolerated well by most men; however, the incidence of adverse events is higher than with either therapy alone. In patients with improved LUTS following combination therapy, the aim of this study is based on the hypothesis that the withdrawal of either therapy will not increase the risk of LUTS aggravation while improving the quality of life.

The investigators plan a prospective, randomized, open-label, parallel trial, comparing alpha-blocker withdrawal and 5-ARI withdrawal to continued combination therapy. Treatments will be allocated in a 1:1:1 ratio, based on IPSS score (≤30% decrease from baseline) and prostate volume (≤35% decrease from baseline).

ELIGIBILITY:
Inclusion Criteria:

* Men aged ≥50 or <80 years AND
* On combination therapy (alpha-blocker and 5-ARI) ≥12 months AND
* IPSS score (≤30% decrease from baseline) AND
* Prostate volume (≤35% decrease from baseline)

Exclusion Criteria:

* Suspected prostate cancer (PSA density >0.15 ng/ml/cc) requiring specific management
* On-going prostatitis or urinary retention
* Acontractile detrusor
* Neurogenic lower urinary tract dysfunction
* Urethral stenosis
* Patient unable or unwilling to provide written informed consent

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-12-08 (Actual); Primary Completion 2023-12-07 (Estimated); Study Completion 2023-12-07 (Estimated)

PRIMARY OUTCOMES:
Change in International Prostate Symptom Score (IPSS) score from baseline | 18 months
  IPSS is the sum of the seven questions with each score ranging from 0 (best) to 5 (worst). IPSS is self-administered at screening and each time-point of month 3, 6, 12, and 18. Seven questions included are incomplete emptying, frequency, intermittency, urgency, weak stream, straining and nocturia. The total IPSS score can range from 0-35 with severity catagories of mild (0 to 7), moderate (8 to 19) or severe (20 to 35). Month 18 is the primary timepoint and earlier timepoints are considered secondary. Change from baseline defined as difference between post-baseline value and baseline value.

SECONDARY OUTCOMES:
Number of adverse events | 3, 6, 12, 18 months
  Adverse events includes; dizziness, headache, pounding heartbeat, weakness. decreased sexual desire, impotence, ejaculatory disorder, gynecomastia, depression, and anxiety.
Change in International Prostate Symptom Score (IPSS) from baseline | 3, 6, 12 months
  IPSS is the sum of the seven questions with each score ranging from 0 (best) to 5 (worst). IPSS is self-administered at screening and each time-point of month 3, 6, and 12. Seven questions included are incomplete emptying, frequency, intermittency, urgency, weak stream, straining and nocturia. The total IPSS score can range from 0-35 with severity catagories of mild (0 to 7), moderate (8 to 19) or severe (20 to 35). Change from baseline defined as difference between post-baseline value and baseline value.
Change in Overactive bladder symptom score (OABSS) from baseline | 3, 6, 12, 18 months
  The OABSS is a symptom assessment questionnaire designed to quantify OAB symptoms into a single score. The questionnaire consists of 4 questions on OAB symptoms with maximum scores ranging from 2 to 5: daytime frequency (2 points), night-time frequency (3 points), urgency (5 points), and UUI (5 points). OABSS is self-administered at screening and each time-point of month 3, 6, 12 and 18. Change from baseline defined as difference between post-baseline value and baseline value.
Change in EuroQol five dimension scale (EQ-5D) score from baseline | 3, 6, 12, 18 months
  The EuroQol five dimension descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The EQ-5D is self-administered at screening and each time-point of month 3, 6, 12 and 18. Change from baseline defined as difference between post-baseline value and baseline value.
Change in Qmax from baseline | 3, 12, 18 months
  The measurement of maximum urinary flow rate (Qmax) is widely used in the assessment of men complaining of lower urinary tract symptoms. Qmax is performed at screening and each time-point of month 3, 12, and 18. Change from baseline defined as difference between post-baseline value and baseline value.
Change in prostate volume from baseline | 18 months
  The measurement of prostate volume is performed at screening and at month 18. Change from baseline defined as difference between post-baseline value and baseline value.
Change in prostate-specific antigen (PSA) level from baseline | 18 months
  The measurement of prostate-specific antigen (PSA) level is performed at screening and at month 18. Change from baseline defined as difference between post-baseline value and baseline value.

CONTACTS AND LOCATIONS:
Overall Officials: Kyo Chul Koo, MD, PhD, Principal Investigator — Yonsei University
Locations (1):
- Gangnam Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Barkin J, Guimaraes M, Jacobi G, Pushkar D, Taylor S, van Vierssen Trip OB. Alpha-blocker therapy can be withdrawn in the majority of men following initial combination therapy with the dual 5alpha-reductase inhibitor dutasteride. Eur Urol. 2003 Oct;44(4):461-6. doi: 10.1016/s0302-2838(03)00367-1. PMID 14499682
- [Result] Nickel JC, Barkin J, Koch C, Dupont C, Elhilali M. Finasteride monotherapy maintains stable lower urinary tract symptoms in men with benign prostatic hyperplasia following cessation of alpha blockers. Can Urol Assoc J. 2008 Feb;2(1):16-21. doi: 10.5489/cuaj.520. PMID 18542722
- See also: Finasteride monotherapy maintains stable lower urinary tract symptoms in men with benign prostatic hyperplasia following cessation of alpha blockers — https://pubmed.ncbi.nlm.nih.gov/18542722/
- See also: Alpha-blocker therapy can be withdrawn in the majority of men following initial combination therapy with the dual 5alpha-reductase inhibitor dutasteride — https://pubmed.ncbi.nlm.nih.gov/14499682/